CLINICAL TRIAL: NCT04657614
Title: The Effect of Alternative Prosthetic Alignments on Sit-to-Stand Proficiency in Transtibial Amputees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Michael Davidson, Assistant Professor Orthotics and Prosthetics, Loma Linda University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 5200455
Record Dates: First submitted 2020-12-01; First posted 2020-12-08 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: Amputation Balance Prosthesis

STUDY DESIGN:
Who Masked: Participant
Masking Description: A sock will be placed over the prosthesis in order for the participant to not know which alignment is used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Neutral Alignment Group (Experimental): A straight pylon with the ankle at neutral.
  Interventions: Other: Neutral Alignment
- Anterior Alignment Group (Experimental): An anteriorly displaced pylon with ankle dorsiflexion at 5 degrees.
  Interventions: Other: Anterior Alignment
- Posterior Alignment Group (Experimental): A posteriorly displaced pylon with 5 degrees of plantarflexion at the ankle.
  Interventions: Other: Posterior Alignment

INTERVENTIONS:
Other: Neutral Alignment — Alignment that is a neutral replicate of the participants prescribed prosthesis.
  Arms: Neutral Alignment Group
Other: Anterior Alignment — Alignment that is anterior displaced pylon.
  Arms: Anterior Alignment Group
Other: Posterior Alignment — Alignment that is posteriorly displaced pylon.
  Arms: Posterior Alignment Group

SUMMARY:
The purpose of this graduate student research study is to determine the effect of various linear and angular prosthetic alignments on K1-K3 unilateral or bilateral TT amputees, as well as test for proficiency, comfort, balance, heart rate and fit during sit to stands.

DETAILED DESCRIPTION:
Initial Visit:

1. Informed consent
2. HIPAA
3. Foot Inspection
4. Review expectations
5. Take measurements
6. Casting

Second Visit: Fitting and adjusting accordingly.

* One person will conduct all the measurements, casting, check sockets, etc. to evade inconsistencies in data collection.
* Begin conducting practice runs on Balance Master at LLU-East Campus.

Third, Fourth and Fifth Visit: Testing (5-10-minute rest period in between each test) *Testing will be video recorded for re-assessment of subjects*

1. Five times sit-to-stand test (5XSTS).
2. Activities-Specific Balance Confidence (ABC-16) scale
3. Balance Master:

   Weight Bearing Squat (WBS) Unilateral Stance (US) Sensory Organization Test (SOT) modified Clinical Test of Sensory Interaction on Balance (mCTSIB) Limits of Stability (LOS)
4. A Polar H10 heart rate monitor will be worn while subjects perform each of the various tests.

ELIGIBILITY:
Inclusion Criteria:

Male and Female below knee amputees (bi-lateral or unilateral)

* 18-70 years of age
* K1-K3 (K-levels/activity levels)

  * K1=patient has the ability or potential to use a prosthesis for transfers or walking on level surfaces at a fixed speed (typical limited or unlimited household ambulator).
  * K2=patient has the ability or potential for walking with the ability to traverse most low-level environmental barriers such as curbs, stairs, or uneven surfaces (typical community ambulator).
  * K3=patient has the ability or potential for walking with variable speed. Has the ability to traverse most environmental barriers and may have vocational, exercise, or recreational activities that demand prosthetic use beyond simple locomotion.
* Those who wear a prosthesis daily for the purpose of walking
* Able to get in and out of a chair
* Prosthetic foot that has the same functional components as the subject's current one

Exclusion Criteria:

Amputation at birth

* Foot amputation at ankle
* Uncontrolled edema in leg compartments
* Compromised skin of the residual limb
* Patients that are 3 months or less post-amputation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2021-07-08 (Actual); Study Completion 2021-07-08 (Actual)

PRIMARY OUTCOMES:
5 Time Sit to Stand Test | three weeks
  The sit to stand test will be administered five times uninterrupted. The participants will sit in a chair and stand up preferably unassisted by researchers. They will be timed.

SECONDARY OUTCOMES:
Activities-Specific Balance Confidence Questionnaire | three weeks
  Measure of balance and confidence in performing various activities.
Balance test | three weeks
  Smart Balance Master system will be used to measure balance and prosthetic alignment during balance test such as limits of stability and weight bearing squat.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Davidson, MSE MPH, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University, Loma Linda, California, United States